CLINICAL TRIAL: NCT05181943
Title: EFFECTIVNESS OF PHOTO BIO-MODULATION IN THE TREATMENT OF CHEMOTHERAPY INDUCED ORAL MUCOSITIS IN CHILDREN WITH ACUTE LEUKEMIA Randomized Controlled Clinical Trial
Brief Title: Effectiveness of Photo-biomodulation in the Treatment of Chemotherapy Induced Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Farida Reayd, Instructor of Oral Medicine, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 332021
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Mucositis
Keywords: mucositis - leukemia - chemotherapy
MeSH Terms: conditions — Mucositis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser irradiation (Test group) (Experimental): laser irradiation over lesion
  Interventions: Device: Simpler diode laser
- Conventional treatment (Control group (Active Comparator)
  Interventions: Drug: Conventional symptomatic treatment

INTERVENTIONS:
Device: Simpler diode laser — Non-contacting irradiation for 30 seconds on three intraoral sites repeated four times
  Arms: Laser irradiation (Test group)
Drug: Conventional symptomatic treatment — Conventional treatment using oracure, BBC spray, miconaz three times daily
  Arms: Conventional treatment (Control group

SUMMARY:
The aim of the current study was to study the effect of diode laser in the treatment of chemotherapy induced mucositis in young patients suffering from leukemia

ELIGIBILITY:
Inclusion Criteria:

* children diagnosed with mucositis and receiving chemotherapy

Exclusion Criteria:

* diabetes
* trismus

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Self-reported pain level | up to 2 weeks
  Participants were asked to report the degree of pain. This was assessed using the visual analogue scale (VAS) which ranges from zero (lowest score) to 10 (highest score). Higher scores indicate higher pain level.
Oral mucositis lesion size | up to 2 weeks
  This was assessed using the World Health Organization oral mucositis lesion score Grade 0: no oral mucositis. Grade1: Presence of soreness and erythema. Grade 2: Presence of painful erythema and ulcerations that do not affect the patient solid food intake.
  Grade3: Confluent ulceration that affect the solid food intake and require liquid diet.
  Grade 4: The patient requires parenteral nutrition.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No